CLINICAL TRIAL: NCT05072015
Title: Systematic Follow up of Second Line Treatments for Parkinson's Disease (Deep Brain Stimulation, Apomorphin Pump, Duodopa Pump)
Acronym: TeSLa-PD
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8355
Record Dates: First submitted 2021-09-30; First posted 2021-10-08 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary purpose: Fluctuations and dyskinesia evolution in Parkinson's disease patients, one year after initiation of deep brain stimulation, apomorphin pump or duodopa pump

Secundary purposes:

* Motor complications evolution at 6 months, 2 and 3 years
* MDS UPDRS III score at 6 months, 1, 2 and 3 years
* non motor complications evolution at 6 months, 1, 2 and 3 years
* cognition and psychiatric complications evolution at 6 months, 1, 2 and 3 years
* cutaneous and digestive complications at 6 months, 1, 2 and 3 years
* neuropathy occurrence at 6 months, 1, 2 and 3 years
* medical treatment and Levodopa equivalent dose modifications at 6 months, 1, 2 and 3 years

ELIGIBILITY:
Inclusion criteria:

* Parkinson disease (UKPDSSB criteria)
* Patient with fluctuations and/or dyskinesia , who need treatment with deep brain stimulation, apomorphin pump or duodopa pump
* MOCA >20
* patient >21 years of age
* patient who has signed protocol acceptation

Exclusion criteria:

* patient who did not give his acceptation for the protocol
* patient with another parkinsonian syndrome than Parkinson' s disease
* MOCA<20
* Patient who does not need second line treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced Parkinson' s disease who need second line treatment
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
MDS UPDRS IV (Movement Disorder Society - Unified Parkin-son Disease Rating Scale) score improvement | 1 year
  Evaluate the evolution of motor fluctuations and dyskinesias at one year in patients. treated with one of the 3 TSLs (bilateral stimulation of the subthalamic nucleus, apomorphine pump and duodopa pump. the higher the score, the more the disease is installed

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu ANHEIM, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Mathieu ANHEIM, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided